CLINICAL TRIAL: NCT05474144
Title: A Two-arm, Double-blind, Randomized, Placebo-controlled Trial Investigating the Efficacy of the Probiotic Dietary Supplement SmartProbio C in the Supportive Supplementation of Patients With a Complicated Course of COVID-19 Infection
Brief Title: Monitoring the Efficacy of a Probiotic Dietary Supplement SmartProbio C in Patients With Severe COVID-19 Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medi Pharma Vision (Industry)
Collaborators: Veterinary Research Institute (Unknown); Brno University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 123666
Record Dates: First submitted 2022-07-21; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: COVID-19
Keywords: COVID-19; probiotics; probiotic supplementation
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum (Experimental): Patients received probiotic supplement SmartProbio C, one capsule twice a day - mornings and evenings before meal - for a period of 2 weeks.
  Interventions: Dietary Supplement: SmartProbio C
- Placebo (Placebo Comparator): Patients received placebo consisting of purified maltodextrin, one capsule twice a day - mornings and evenings before meal - for a period of 2 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: SmartProbio C — Probiotic supplement consisting of 19 strains (Lactobacillus acidophilus NCFM, Bifidobacterium lactis, subsp. Infantis Bi-07, Lactobacillus rhamnosus LR22, Lactobacillus acidophilus LA14, Lactobacillus rhamnosus LGG, Bifidobacterium lactis HN019, Bifidobacterium lactis Bl-04, Lactobacillus acidophilus LA 11 ONLLY, Lactobacillus rhamnosus HN001, Lactobacillus plantarum LP ONLLY, Lactobacillus casei LC18, Bifidobacterium breve BB8, Lactobacillus reuteri LE16, Bifidobacterium lactis BI516, Streptococcus thermophilus ST6, Bifidobacterium animalis BA77, Bifidobacterium bifidum BB47, Bifidobacterium longum BL88 ONLLY, Bifidobacterium infantis BI211) in different ratios. Probiotic mixture enclosed in HPMC (hydroxypropylmethylcelulose) capsule, 25 billion CFU (colony-forming units) in each capsule. As a filling agent mix of inulin and maltodextrin was used. Dosage twice a day.
  Arms: Verum
Dietary Supplement: Placebo — Placebo. HPMC (hydroxypropylmethylcelulose) capsule filled with maltodextrin. Dosage twice a day.
  Arms: Placebo

SUMMARY:
The aim of the study is to test the efficacy of the probiotic SmartProbio C in patients with a severe course of COVID-19 infection. Patients were randomly divided into two arms between the probiotic group and the placebo group. They were further divided into four groups according to 1) BMI (Body mass index; <=30/>30), 2) age (<=65/>65), 3) CRP (C-reactive protein; <=100/>100), 4) chronic lung disease (yes/no). Gut microbiome analysis and its changes in selected parameters (amount of lactobacilli, bifidobacteria, Akkermansia, Proteobacteria, Firmicutes/Bacteroidetes ratio) were chosen as the primary endpoint. Other assessed indicators include:

* Tracking of time to clinical improvement by two points on a seven-point ordinal scale for clinical improvement according to R&D Blueprint: COVID-19 Therapeutic Trial Synopsis (WHO, 2020) or time to hospital discharge (whichever comes first)
* Monitoring the length of oxygen dependence
* Monitoring of laboratory markers of inflammation - serum peripheral blood CRP levels
* Monitoring of mortality

ELIGIBILITY:
Inclusion Criteria:

* The subject is willing and able to provide informed consent prior to any study procedure.
* Age at the time of screening between 18 and 85 years inclusive.
* Coronavirus (SARS-CoV-2) infection confirmed by polymerase chain reaction (PCR) or immunochromatographic detection of SARS CoV-2 specific antigens no more than three days prior to randomization.
* COVID-19 symptoms lasting less than or equal to seven days, including.
* Subject is currently hospitalized and requires medical care due to COVID-19 disease and was admitted at most two days prior to randomization.
* Peripheral blood oxygen saturation <94% on air (as measured by pulse oximetry or arterial blood sampling) at the time of inclusion in the trial.

Exclusion Criteria:

* Participation in any other clinical trial of an experimental treatment for COVID-19 disease.
* Concomitant treatment of COVID-19 with other non-standard-of-care medications less than 24 hours prior to initiation of the study intervention dosing (excluding remdesivir, corticosteroids, casirivimab, imdevimab, or bamlanivimab).
* Immunosuppressant treatment three months prior to hospital admission (excluding topical and inhaled corticosteroids or systemically administered corticosteroids at a dose equivalent to <40 mg Prednisone)
* Necessity of invasive pulmonary ventilation.
* Patients with known primary or secondary immunodeficiency.
* History of Crohn's disease or ulcerative colitis.
* Abnormal screening laboratory results - laboratory abnormalities that, in the opinion of the investigator, will interfere with completion of participation in the clinical trial or will interfere with the results of the trial.
* Participation in another clinical trial of a drug or medical device, or less than 30 days have elapsed since the completion of participation in another trial or use of the investigational drug or device.
* Other probiotic supplementation.
* Hypersensitivity to any ingredient of a product administered during a clinical trial.
* Women who are pregnant or breastfeeding.
* Patients with preterminal and terminal organ failure (COPD GOLD 3 and 4, CKD G4 and G5, NYHA 3 and 4).
* Any condition that, in the opinion of the investigator, may compromise the patient's ability to provide informed consent and/or comply with all required study procedures.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Gut microbiome | The first sample was taken at the beginning of hospitalization before the start of supplementation, the second at discharge from the hospital, but not later than on the 14th day of hospitalization.
  Changes in selected parameters of gut microbiome (amount of lactobacilli, bifidobacteria, Akkermansia, Proteobacteria, and Firmicutes/Bacteroidetes ratio) were chosen as the primary endpoint.

SECONDARY OUTCOMES:
Length of hospitalisation | From the date of admission to hospital until discharge from hospital or above defined two point improvement, whichever comes first
  Tracking of time to clinical improvement by two points on a seven-point ordinal scale for clinical improvement according to R&D Blueprint: COVID-19 Therapeutic Trial Synopsis (WHO, 2020), or time to hospital discharge (whichever comes first).
Monitoring the length of oxygen dependence | From the beginning of the provision of HFOT (high flow oxygen therapy) to the end of the provision of HFOT
  Measurement of the time it was necessary to provide HFOT (high flow oxygen therapy) to the patient
CRP (C-reactive protein) monitoring | On the first day of admission to hospital and on the day of hospital discharge, but no later than 14th day
  Monitoring of laboratory marker of inflammation - serum peripheral blood CRP levels
Monitoring mortality rates | From the date of admission to hospital until discharge from hospital or death, whichever comes first
  The percentage of deaths in the placebo group compared to percentage of deaths in the verum group

CONTACTS AND LOCATIONS:
Overall Officials: Petr Rysavka, Ph.D., Principal Investigator — Medi Pharma Vision
Locations (2):
- Czechia (2):
  - Medi Pharma Vision, Brno
  - Brno University Hospital, Brno

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adler Sorensen C, Fuglsang E, Jorgensen CS, Laursen RP, Larnkjaer A, Molgaard C, Ritz C, Michaelsen KF, Krogfelt KA, Frokiaer H. Probiotics and the immunological response to infant vaccinations; a double-blind randomized controlled trial. Clin Microbiol Infect. 2019 Apr;25(4):511.e1-511.e7. doi: 10.1016/j.cmi.2018.07.031. Epub 2018 Aug 9. PMID 30099133
- [Background] Baud D, Dimopoulou Agri V, Gibson GR, Reid G, Giannoni E. Using Probiotics to Flatten the Curve of Coronavirus Disease COVID-2019 Pandemic. Front Public Health. 2020 May 8;8:186. doi: 10.3389/fpubh.2020.00186. eCollection 2020. No abstract available. PMID 32574290
- [Background] Bottari B, Castellone V, Neviani E. Probiotics and Covid-19. Int J Food Sci Nutr. 2021 May;72(3):293-299. doi: 10.1080/09637486.2020.1807475. Epub 2020 Aug 12. PMID 32787470
- [Background] Doron S, Snydman DR. Risk and safety of probiotics. Clin Infect Dis. 2015 May 15;60 Suppl 2(Suppl 2):S129-34. doi: 10.1093/cid/civ085. PMID 25922398
- [Background] Li KJ, Chen ZL, Huang Y, Zhang R, Luan XQ, Lei TT, Chen L. Dysbiosis of lower respiratory tract microbiome are associated with inflammation and microbial function variety. Respir Res. 2019 Dec 3;20(1):272. doi: 10.1186/s12931-019-1246-0. PMID 31796027
- [Background] Xu K, Cai H, Shen Y, Ni Q, Chen Y, Hu S, Li J, Wang H, Yu L, Huang H, Qiu Y, Wei G, Fang Q, Zhou J, Sheng J, Liang T, Li L. [Management of COVID-19: the Zhejiang experience]. Zhejiang Da Xue Xue Bao Yi Xue Ban. 2020 Feb 21;49(2):147-157. doi: 10.3785/j.issn.1008-9292.2020.02.02. Chinese. PMID 32391658
- [Background] Nguyen QV, Chong LC, Hor YY, Lew LC, Rather IA, Choi SB. Role of Probiotics in the Management of COVID-19: A Computational Perspective. Nutrients. 2022 Jan 10;14(2):274. doi: 10.3390/nu14020274. PMID 35057455